CLINICAL TRIAL: NCT03280082
Title: Operational Experience for the Use of the Mid-Upper Arm Circumference (MUAC) as the Basic Criterion for Admission, Follow-up and Exit of the Ambulatory Nutrition Program in Two CRENAS, Madaoua District, Niger
Brief Title: Use of MUAC as Basic Criterion for Admission, Follow-up and Exit From the Ambulatory Nutrition Program
Acronym: MUAC120
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Spain (Other); Direction de la Nutrition du Niger (Unknown); District Sanitaire de Madaoua, Niger (Unknown); Direction Régionale Sanitaire de Tahoua, Niger (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUAC 120
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MUAC Program (Other): At the CRENAS, MUAC as unique anthropometric criteria for admission, monitoring, and care for the SAM output will be used.
  The criteria for admission include:
  * MUAC <120 mm
  * Bilateral edema of grade + or ++
  The criteria for release of care include:
  * MUAC ≥ 125 mm at 2 consecutive visits
  * Minimum stay 3 weeks in the program
  * Absence of acute medical complications
  * Absence of edema
  Interventions: Other: MUAC Program
- Standard Program (Other): Regular screenings in the communities on children between 6 and 59 months of age. Children with MUAC<125 mm will be referred to Nutrition Centers for admission.
  The criteria for admission include:
  * MUAC<115 mm and/or
  * Z score <-3 and /or
  * Bilateral edema of grade + or ++
  The criteria for release of care include:
  * MUAC ≥ 125 mm at 2 consecutive visits
  * Minimum stay 3 weeks in the program
  * Absence of acute medical complications
  * Absence of edema
  Interventions: Other: Standard Program

INTERVENTIONS:
Other: MUAC Program — All children admitted to the PB program will receive standard care according to the national Protocol and that of MSF, including preventive and therapeutic care at admission as well as hospital care in case of clinical complications. There will be no change in the Protocol for the hospital care to the CRENI (Center of Intensive Nutritional Rehabilitation). RUTF (Ready-to-Use therapeutic food) will be distributed on a weekly basis according to the dosage of RUTF in the national protocol.
  Arms: MUAC Program
Other: Standard Program — All children admitted to the standard program will receive standard care according to national and MSF protocols, including preventive and therapeutic care on admission as well as hospital care in case of clinical complications. RUTF will be distributed on a weekly basis according to the dosage of RUTF in the national protocol.
  Arms: Standard Program

SUMMARY:
The aim of this study is to provide comprehensive documentation of the relevant results and operational implications of this new model using Mid-Upper Arm Circumference (MUAC) as the single anthropometric criterion for admission, monitoring and exit of non- complicated in Niger.

DETAILED DESCRIPTION:
This is a first operational experiment using Mid-Upper Arm Circumference (MUAC) as the single anthropometric criterion for the admission, monitoring and exit of the management of uncomplicated SAM (Severe Acute Malnutrition) in Niger, specific data as well as data from routine program will be collected to allow comprehensive documentation of all relevant results and operational implications of this new model. The experiment based on the use of the single anthropometric threshold for admission of a Mid-Upper Arm Circumference (MUAC)<120 mm, which includes both children currently classified as having SAM (currently with PB <115 mm) and acute malnutrition moderate (MAM, currently with a Mid-Upper Arm Circumference (MUAC)<125 mm), as well as a follow-up of children with a Mid-Upper Arm Circumference (MUAC)≥ 120 mm, will identify how children respond to treatment and benefit of the spectrum of acute malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted for non-complicated SAM (Severe Acute Malnutrition) treatment

Exclusion Criteria:

* Children between the ages of 6 and 59 months who were recently excluded from treatment by admission criteria based on MUAC (Sabon Guida site) but were previously eligible for treatment (ie MUAC ≥ 120 and Z score <-3).

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6200 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Nutritional recovery | 18 months
  Compare the average daily weight gain and the duration of the nutritional treatment per group compare the results of the PB programme, including the overall risk of recovery, transfer, of abandonment, of death, of PB and weight gain and the length of stay by age (6-23 months, compared to 24-59 months), compared the results of the program standard;

SECONDARY OUTCOMES:
Readmission risks | 3 months
  Assessment of the risk of readmission 3 months after discharged of the child will be evaluated at 3 months (+/- one week) after discharged of the child
Deaths | 18 months
  Compare the death rate between the two groups

OTHER OUTCOMES:
Documentation of the results | 18 months
  Document coverage of the nutrition program before and after the implementation of the

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca GRAIS, PhD, Study Director — Epicentre
Locations (1):
- CRENAS, Madaoua, Niger

REFERENCES:
- [Derived] Isanaka S, Hedt-Gauthier BL, Grais RF, Allen BGS. Estimating program coverage in the treatment of severe acute malnutrition: a comparative analysis of the validity and operational feasibility of two methods. Popul Health Metr. 2018 Jul 3;16(1):11. doi: 10.1186/s12963-018-0167-3. PMID 29970172